CLINICAL TRIAL: NCT00291486
Title: Phase I Trial of Oral Capecitabine Combined With 131I-huA33 in Patients With Metastatic Colorectal Cancer
Brief Title: Capecitabine and 131I-huA33 in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LUD2002-017; R21CA108145-01A1 (NIH)
Record Dates: First submitted 2006-02-10; First posted 2006-02-14 (Estimated); Results first posted 2022-01-11 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): 20 millicurie (mCi) 131I-huA33, 1500 mg/m2/day capecitabine
  All patients received an initial dose of 5 mg huA33 conjugated to 5-8 mCi 131I on day 0.
  This was followed 7 ± 2 days later by inpatient administration of a single infusion of 131I-huA33 with a constant protein dose of 10 mg/m2 huA33.
  Capecitabine was administered in 2 divided doses per day on days 1-14 of each 21-day cycle for a total of 4 cycles. Daily doses were rounded to the nearest 150 mg.
  Interventions: Drug: Capecitabine; Drug: 131I-huA33 (131-Iodine on humanised monoclonal antibody A33)
- Cohort 2 (Experimental): 30 millicurie (mCi) 131I-huA33, 1500 mg/m2/day capecitabine
  All patients received an initial dose of 5 mg huA33 conjugated to 5-8 mCi 131I on day 0.
  This was followed 7 ± 2 days later by inpatient administration of a single infusion of 131I-huA33 with a constant protein dose of 10 mg/m2 huA33.
  Capecitabine was administered in 2 divided doses per day on days 1-14 of each 21-day cycle for a total of 4 cycles. Daily doses were rounded to the nearest 150 mg.
  Interventions: Drug: Capecitabine; Drug: 131I-huA33 (131-Iodine on humanised monoclonal antibody A33)
- Cohort 3 (Experimental): 30 millicurie (mCi) 131I-huA33, 1000 mg/m2/day capecitabine
  All patients received an initial dose of 5 mg huA33 conjugated to 5-8 mCi 131I on day 0.
  This was followed 7 ± 2 days later by inpatient administration of a single infusion of 131I-huA33 with a constant protein dose of 10 mg/m2 huA33.
  Capecitabine was administered in 2 divided doses per day on days 1-14 of each 21-day cycle for a total of 4 cycles. Daily doses were rounded to the nearest 150 mg.
  Interventions: Drug: Capecitabine; Drug: 131I-huA33 (131-Iodine on humanised monoclonal antibody A33)
- Cohort 4 (Experimental): 40 millicurie (mCi) 131I-huA33, 1000 mg/m2/day capecitabine
  All patients received an initial dose of 5 mg huA33 conjugated to 5-8 mCi 131I on day 0.
  This was followed 7 ± 2 days later by inpatient administration of a single infusion of 131I-huA33 with a constant protein dose of 10 mg/m2 huA33.
  Capecitabine was administered in 2 divided doses per day on days 1-14 of each 21-day cycle for a total of 4 cycles. Daily doses were rounded to the nearest 150 mg.
  Interventions: Drug: Capecitabine; Drug: 131I-huA33 (131-Iodine on humanised monoclonal antibody A33)
- Cohort 5 (Experimental): 40 millicurie (mCi) 131I-huA33, 1250 mg/m2/day capecitabine
  All patients received an initial dose of 5 mg huA33 conjugated to 5-8 mCi 131I on day 0.
  This was followed 7 ± 2 days later by inpatient administration of a single infusion of 131I-huA33 with a constant protein dose of 10 mg/m2 huA33.
  Capecitabine was administered in 2 divided doses per day on days 1-14 of each 21-day cycle for a total of 4 cycles. Daily doses were rounded to the nearest 150 mg.
  Interventions: Drug: Capecitabine; Drug: 131I-huA33 (131-Iodine on humanised monoclonal antibody A33)

INTERVENTIONS:
Drug: Capecitabine — Capecitabine was administered orally at doses between 1000 and 1500 mg/m2/day depending on assigned dose level for 14 days per 21-day cycle. Daily doses were rounded to the nearest 150 mg.
  Other Names: Xeloda
Drug: 131I-huA33 (131-Iodine on humanised monoclonal antibody A33) — All patients received a dose of 5 mg huA33 conjugated to 5-8 mCi 131I. The therapy dose of 131I-huA33 comprised a constant protein dose of 10 mg/m2 huA33 regardless of dose level. The 131I-huA33 therapy dose was determined by the assigned dose level (i.e. 20, 30 or 40 mCi/m2 131I).

SUMMARY:
The purpose of this clinical trial is to determine whether it is safe to treat patients with advanced colorectal cancer, with humanised A33 antibody tagged with radioactive iodine (131I-huA33) in combination with chemotherapy (capecitabine).

DETAILED DESCRIPTION:
This clinical trial tests the combination of humanised A33 monoclonal antibody tagged with radioactive iodine 131 (131I-huA33) together with capecitabine chemotherapy in patients with advanced colorectal cancer.

When colorectal cancer has spread to other organs, it is generally considered incurable but with a limited number of treatment options. Colorectal cancer cells express proteins on their surface known as antigens, and one of these is called the A33 antigen. An antibody which targets the A33 antigen was initially developed in the mouse and found to bind to human colorectal cancer cells. Because humans developed immune reactions when given the mouse antibody, an antibody, which is more like normal human antibodies, was developed (humanised A33 antibody). In order to increase its effectiveness, radioactive iodine (131I) has been attached to the antibody so that the antibody can deliver radiation directly to colorectal cancer cells. Previous studies have shown that both the unlabelled humanised A33 antibody as well as the humanised A33 antibody tagged with radioactive iodine can be administered safely to humans with no major allergic reactions. The addition of chemotherapy to radiolabelled 131I-huA33 may result in a treatment that is more effective for the treatment of colorectal cancer than either agent alone.

The purpose of this study is to determine whether it is safe to give humanised A33 antibody tagged with radioactive iodine together with chemotherapy. Different dose levels of radioactive iodine attached to a constant dose of antibody will be given together with a fixed total daily capecitabine chemotherapy dose. Providing humanised A33 antibody tagged with radioactive iodine and chemotherapy is tolerated well without major side effects, the dose of capecitabine chemotherapy given with 131I-huA33 will also be increased in order to determine the highest dose that can be given safely in combination with radio-labelled 131I-huA33. The effectiveness of the treatment combination against advanced colorectal cancer will also be assessed.

Patients with advanced colorectal cancer who have never previously received chemotherapy using capecitabine may be eligible to participate in the study. A total of between 15 and 30 patients are expected to be recruited.

Screening blood tests will be performed to determine eligibility, as well as baseline heart and lung function tests and appropriate scans to measure tumour size and assess radiation within the body. Patients will be given a trace-labelled (small radiation dose) infusion of 131I-huA33 into a vein followed a week later by the treatment infusion of 131I-huA33. The first infusion will be given as an outpatient, but for the second, patients will be hospitalized and confined to a radiation-shielded room until radiation levels fall to safe limits. Oral iodine drops will also be given for 28 days in order to protect the thyroid gland from the effects of radioactive iodine. Capecitabine chemotherapy will be taken orally and will commence at the time of the treatment infusion. Each cycle of capecitabine chemotherapy involves the medication being taken twice per day for a total of 14 days followed by 7 days rest. A total of 4 cycles of capecitabine will be given after the treatment infusion.

Blood samples will be taken just before the treatment infusion and then weekly for 13 weeks. There will be weekly physical examinations until 9 weeks after the treatment infusion and again at 12 weeks. Total study duration is 13 weeks from the trace-labelled infusion of 131I-huA33, that is 12 weeks from the treatment infusion of 131I-huA33. Patients will only receive one treatment infusion of 131I-huA33 antibody.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic colorectal cancer.
* Histologically or cytologically proven colorectal cancer.
* Measurable disease on CT scan with at least one lesion >/= 2cm diameter (to allow adequate infusion imaging).
* Expected survival of at least 4 months.
* ECOG performance status 0-2.
* Vital laboratory parameters should be within normal range including:

  1. Neutrophils >/= 1.5 x 10^9/L;
  2. Platelets >/= 150 x 10^9/L;
  3. Serum bilirubin </= 34 micromol/L;
  4. Calculated creatinine clearance > 50 ml/min.
* Age >/= 18 years.
* Able and willing to give valid written informed consent.

Exclusion Criteria:

* Previous treatment with capecitabine.
* Untreated active metastatic disease to the central nervous system (new or enlarging lesions on CT or MRI), or within 3 months of treatment (ie surgery or radiotherapy) for brain metastases.
* Other serious illnesses, eg, serious infections requiring antibiotics, bleeding disorders.
* Liver involvement with metastatic disease > 50% liver volume.
* Chemotherapy, radiation therapy, or immunotherapy within 4 weeks before study entry (6 weeks for nitrosoureas).
* Previous external beam irradiation except if: (i) it was for standard adjuvant pelvic radiation for rectal cancer; (ii) it was for localised irradiation for skin cancer; or (iii) the sum total of all previous external beam irradiation port areas is not greater than 25% of the total red marrow.
* Previous treatment with a monoclonal antibody or antibody fragment AND a positive huA33 human anti-human antibody (HAHA) titre.
* Concomitant treatment with systemic corticosteroids. Topical or inhalational corticosteroids are permitted.
* Mental impairment that may compromise the ability to give informed consent and comply with the requirements of the study.
* Lack of availability of the patient for clinical and laboratory follow-up assessment.
* Participation in any other clinical trial involving another investigational agent within 4 weeks prior to enrollment.
* Pregnancy or breastfeeding.
* Women of childbearing potential: Refusal or inability to use effective means of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2003-10 (Actual); Primary Completion 2008-01-03 (Actual); Study Completion 2012-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Andrew M Scott, MBBS, DDU MD, Principal Investigator — Ludwig Institute for Cancer Research
Locations (1):
- Ludwig Institute Oncology Unit and Tumor Targeting Program, Austin Health, Heidelberg, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437
- [Result] Herbertson RA, Tebbutt NC, Lee FT, Gill S, Chappell B, Cavicchiolo T, Saunder T, O'Keefe GJ, Poon A, Lee ST, Murphy R, Hopkins W, Scott FE, Scott AM. Targeted chemoradiation in metastatic colorectal cancer: a phase I trial of 131I-huA33 with concurrent capecitabine. J Nucl Med. 2014 Apr;55(4):534-9. doi: 10.2967/jnumed.113.132761. Epub 2014 Feb 20. PMID 24556590

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: 20 millicurie (mCi) 131I-huA33, 1500 mg/m2/day capecitabine
  All patients received an initial dose of 5 mg huA33 conjugated to 5-8 mCi 131I on day 0.
  This was followed 7 ± 2 days later by inpatient administration of the therapy dose given as a single infusion of 131I-huA33 with a constant protein dose of 10 mg/m2 huA33. The 131I-huA33 therapy dose was determined by the assigned dose level (i.e. 20, 30 or 40 mCi/m2 131I).
  Capecitabine was administered at doses between 1000 and 1500 mg/m2/day depending on assigned dose level for 14 days per 21-day cycle for 4 cycles. Daily doses were rounded to the nearest 150 mg.
- Cohort 2: 30 millicurie (mCi) 131I-huA33, 1500 mg/m2/day capecitabine
  All patients received an initial dose of 5 mg huA33 conjugated to 5-8 mCi 131I on day 0.
  This was followed 7 ± 2 days later by inpatient administration of the therapy dose given as a single infusion of 131I-huA33 with a constant protein dose of 10 mg/m2 huA33. The 131I-huA33 therapy dose was determined by the assigned dose level (i.e. 20, 30 or 40 mCi/m2 131I).
  Capecitabine was administered at doses between 1000 and 1500 mg/m2/day depending on assigned dose level for 14 days per 21-day cycle for 4 cycles. Daily doses were rounded to the nearest 150 mg.
- Cohort 3: 30 millicurie (mCi) 131I-huA33, 1000 mg/m2/day capecitabine
  All patients received an initial dose of 5 mg huA33 conjugated to 5-8 mCi 131I on day 0.
  This was followed 7 ± 2 days later by inpatient administration of the therapy dose given as a single infusion of 131I-huA33 with a constant protein dose of 10 mg/m2 huA33. The 131I-huA33 therapy dose was determined by the assigned dose level (i.e. 20, 30 or 40 mCi/m2 131I).
  Capecitabine was administered at doses between 1000 and 1500 mg/m2/day depending on assigned dose level for 14 days per 21-day cycle for 4 cycles. Daily doses were rounded to the nearest 150 mg.
- Cohort 4: 40 millicurie (mCi) 131I-huA33, 1000 mg/m2/day capecitabine
  All patients received an initial dose of 5 mg huA33 conjugated to 5-8 mCi 131I on day 0.
  This was followed 7 ± 2 days later by inpatient administration of the therapy dose given as a single infusion of 131I-huA33 with a constant protein dose of 10 mg/m2 huA33. The 131I-huA33 therapy dose was determined by the assigned dose level (i.e. 20, 30 or 40 mCi/m2 131I).
  Capecitabine was administered at doses between 1000 and 1500 mg/m2/day depending on assigned dose level for 14 days per 21-day cycle for 4 cycles. Daily doses were rounded to the nearest 150 mg.
- Cohort 5: 40 millicurie (mCi) 131I-huA33, 1250 mg/m2/day capecitabine
  All patients received an initial dose of 5 mg huA33 conjugated to 5-8 mCi 131I on day 0.
  This was followed 7 ± 2 days later by inpatient administration of the therapy dose given as a single infusion of 131I-huA33 with a constant protein dose of 10 mg/m2 huA33. The 131I-huA33 therapy dose was determined by the assigned dose level (i.e. 20, 30 or 40 mCi/m2 131I).
  Capecitabine was administered at doses between 1000 and 1500 mg/m2/day depending on assigned dose level for 14 days per 21-day cycle for 4 cycles. Daily doses were rounded to the nearest 150 mg.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Started | 3 | 6 | 3 | 3 | 4
Completed | 2 | 3 | 2 | 2 | 3
Not Completed | 1 | 3 | 1 | 1 | 1
Not completed — Adverse Event | 0 | 3 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1
Not completed — Disease progression | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: 20 mCi 131I-huA33, 1500 mg/m2/day capecitabine
  All patients received an initial dose of 5 mg huA33 conjugated to 5-8 mCi 131I on day 0.
  This was followed 7 ± 2 days later by inpatient administration of the therapy dose given as a single infusion of 131I-huA33 with a constant protein dose of 10 mg/m2 huA33. The 131I-huA33 therapy dose was determined by the assigned dose level (i.e. 20, 30 or 40 mCi/m2 131I).
  Capecitabine was administered at doses between 1000 and 1500 mg/m2/day depending on assigned dose level for 14 days per 21-day cycle for 4 cycles. Daily doses were rounded to the nearest 150 mg.
- Cohort 2: 30 mCi 131I-huA33, 1500 mg/m2/day capecitabine
  All patients received an initial dose of 5 mg huA33 conjugated to 5-8 mCi 131I on day 0.
  This was followed 7 ± 2 days later by inpatient administration of the therapy dose given as a single infusion of 131I-huA33 with a constant protein dose of 10 mg/m2 huA33. The 131I-huA33 therapy dose was determined by the assigned dose level (i.e. 20, 30 or 40 mCi/m2 131I).
  Capecitabine was administered at doses between 1000 and 1500 mg/m2/day depending on assigned dose level for 14 days per 21-day cycle for 4 cycles. Daily doses were rounded to the nearest 150mg.
- Cohort 3: 30 mCi 131I-huA33, 1000 mg/m2/day capecitabine
  All patients received an initial dose of 5 mg huA33 conjugated to 5-8 mCi 131I on day 0.
  This was followed 7 ± 2 days later by inpatient administration of the therapy dose given as a single infusion of 131I-huA33 with a constant protein dose of 10 mg/m2 huA33. The 131I-huA33 therapy dose was determined by the assigned dose level (i.e. 20, 30 or 40 mCi/m2 131I).
  Capecitabine was administered at doses between 1000 and 1500 mg/m2/day depending on assigned dose level for 14 days per 21-day cycle for 4 cycles. Daily doses were rounded to the nearest 150 mg.
- Cohort 4: 40 mCi 131I-huA33, 1000 mg/m2/day capecitabine
  All patients received an initial dose of 5 mg huA33 conjugated to 5-8 mCi 131I on day 0.
  This was followed 7 ± 2 days later by inpatient administration of the therapy dose given as a single infusion of 131I-huA33 with a constant protein dose of 10 mg/m2 huA33. The 131I-huA33 therapy dose was determined by the assigned dose level (i.e. 20, 30 or 40 mCi/m2 131I).
  Capecitabine was administered at doses between 1000 and 1500 mg/m2/day depending on assigned dose level for 14 days per 21-day cycle for 4 cycles. Daily doses were rounded to the nearest 150 mg.
- Cohort 5: 40 mCi 131I-huA33, 1250 mg/m2/day capecitabine
  All patients received an initial dose of 5 mg huA33 conjugated to 5-8 mCi 131I on day 0.
  This was followed 7 ± 2 days later by inpatient administration of the therapy dose given as a single infusion of 131I-huA33 with a constant protein dose of 10 mg/m2 huA33. The 131I-huA33 therapy dose was determined by the assigned dose level (i.e. 20, 30 or 40 mCi/m2 131I).
  Capecitabine was administered at doses between 1000 and 1500 mg/m2/day depending on assigned dose level for 14 days per 21-day cycle for 4 cycles. Daily doses were rounded to the nearest 150 mg.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Total
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 4 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 3 | 3 | 2 | 13
  >=65 years | 0 | 4 | 0 | 0 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 0 | 1 | 6
  Male | 2 | 4 | 1 | 3 | 3 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 5 | 3 | 3 | 4 | 17
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Australia | 3 | 6 | 3 | 3 | 4 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Dose-Limiting Toxicities (DLT)
Description: Adverse events were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE v3.0). DLT was defined as any of the following related events:
  Any grade 2 or greater allergic reaction related to huA33. Any grade ≥ 3 non-haematological toxicity related to 131I-huA33 or capecitabine.
  * These toxicities included palmar plantar erythema, but skin rash thought to be related to huA33 protein was not a DLT as previous studies have shown no relation of this toxicity to dose of huA33 or radioiodine dose.
  * Capecitabine cardiotoxicity grade ≥ 3 - including vasospasm, acute coronary syndrome and arrhythmia, necessitated the cessation of study drug in the affected patient but were not considered DLT as these are recognized as idiosyncratic in nature and not known to be related to capecitabine dose.
  Any grade ≥ 4 neutropenia ≥ 7 days in duration or any thrombocytopenia with a platelet count < 10 x 10^9/L.
Time Frame: 7 weeks
Population: All patients who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2: 30 mCi 131I-huA33, 1500 mg/m2/day capecitabine
  All patients received an initial dose of 5 mg huA33 conjugated to 5-8 mCi 131I on day 0.
  This was followed 7 ± 2 days later by inpatient administration of the therapy dose given as a single infusion of 131I-huA33 with a constant protein dose of 10 mg/m2 huA33. The 131I-huA33 therapy dose was determined by the assigned dose level (i.e. 20, 30 or 40 mCi/m2 131I).
  Capecitabine was administered at doses between 1000 and 1500 mg/m2/day depending on assigned dose level for 14 days per 21-day cycle for 4 cycles. Daily doses were rounded to the nearest 150 mg.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 4
Participants | 0 | 2 | 0 | 0 | 0

2. Secondary Outcome: Number of Patients With Tumour Response Assessed by Response Evaluation Criteria in Solid Tumors (RECIST).
Description: Tumor responses were evaluated using appropriate imaging and categorized according to RECIST at Screening (within 2 weeks of the first dose of study treatment), and at week 13. Per RECIST, target lesions are categorized as follows: complete response (CR): disappearance of all target lesions; partial response (PR): ≥ 30% decrease in the sum of the longest diameter of target lesions; progressive disease (PD): ≥ 20% increase in the sum of the longest diameter of target lesions; stable disease (SD): small changes that do not meet above criteria (Therasse et al 2000).
Time Frame: 13 weeks
Population: All patients who received at least one dose of study treatment and were evaluable for response. One patient in Cohort 5 was not evaluable due to the patient's request to discontinue the study prior to this evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 3
Participants
  CR | 0 | 0 | 0 | 0 | 0
  PR | 0 | 1 | 0 | 0 | 0
  SD | 1 | 3 | 2 | 1 | 3
  PD | 2 | 2 | 1 | 2 | 0

3. Secondary Outcome: Biodistribution of 131I-huA33 Measured by Whole Body Clearance and Normal Organ Clearance Reported as Mean Biological Half-life (T1/2 Biological) After Initial 131I-huA33 Infusion
Description: T1/2 biological is the clearance of the isotope from the whole body. Following the initial 131I-huA33 infusion, gamma camera scans were acquired over a 1 week period (1-4 hours, Day 1, Day 2 or 3, and Day 4 or 5). Whole body clearance, or biological half time, T1/2 biological, was calculated from the whole body anterior and posterior planar images. A region of interest (ROI) was calculated to encompass the whole body, and for each ROI at each time point, the mean counts per pixel per minute was normalised to imaging time point Day 1.
Time Frame: 1 week
Population: All patients who received the initial infusion of 131I-huA33.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Cohorts 1-5: All patients received an initial dose of 5 mg huA33 conjugated to 5-8 mCi 131I on day 0.
  This was followed 7 ± 2 days later by inpatient administration of the therapy dose given as a single infusion of 131I-huA33 with a constant protein dose of 10 mg/m2 huA33. The 131I-huA33 therapy dose was determined by the assigned dose level (i.e. 20, 30 or 40 mCi/m2 131I).
  Capecitabine was administered at doses between 1000 and 1500 mg/m2/day depending on assigned dose level for 14 days per 21-day cycle for 4 cycles. Daily doses were rounded to the nearest 150 mg.
Arm/Group | Cohorts 1-5
Number analyzed (Participants) | 19
hours
  Whole Body Clearance (T1/2 biologic) | 219.56 (62.81)
  Normal Organ Clearance in the Liver (T1/2 biological - liver) | 62.29 (22.05)
  Normal Organ Clearance in the kidney (T1/2 biological - kidney) | 104.89 (56.22)

4. Secondary Outcome: Mean Specific Absorbed Dose of 131I-huA33 for Normal Organs Calculated From the Initial Infusion
Description: Gamma camera imaging with anterior and posterior whole body scans using conjugate view methodology were performed on four occasions (1-4 hours, Day 1, Day 2 or 3, and Day 4 or 5) following completion of the intravenous initial infusion.
  Dosimetric analysis was performed on the series of gamma camera whole-body planar images acquired in all patients following the first infusion.
  Organ radioactivity content was estimated from the geometric mean of anterior and posterior regions of interest counts. The counts for each organ were corrected for background using regions of interest drawn adjacent to each organ where whole body thickness was comparable.
Time Frame: 1 week
Population: All patients who received the initial infusion of 131I-huA33.
Measure: Mean (Standard Deviation); unit: cGy/MBq
Arm/Group | Cohorts 1-5
Number analyzed (Participants) | 19
cGy/MBq
  Liver | 0.12 (0.03)
  Spleen | 0.18 (0.06)
  Kidney | 0.14 (0.05)
  Lung | 0.09 (0.03)
  Red Marrow | 0.056 (0.011)

5. Secondary Outcome: Mean Total Tumor Dose of 131I-huA33
Description: Gamma camera imaging were performed on four occasions (1-4 hours, Day 1, Day 2 or 3, and Day 4 or 5) following completion of the initial infusion and 7+2 days post-therapy infusion in week 2, and again in week 3 or 4 and week 5 following the therapy infusion.
  Dosimetry analysis was performed on the series of gamma camera whole-body planar images.
  Tumor radioactivity content after the initial infusion was estimated from the geometric mean of anterior and posterior regions of interest counts. The counts for each organ were corrected for background using regions of interest drawn adjacent to each tumor. Resultant counts were converted to activity using a camera sensitivity factor calculated from a gamma camera standard of known activity which was scanned at the same time.
Time Frame: 5 weeks
Population: All patients who received the initial and therapy infusions and had tumors of sufficient size for accurate tumor quantitation and dosimetry. Nine patients had tumors too small to be analyzed. Results are presented by the radiolabeled dose of huA33 given as well as all patients.
Measure: Mean (Standard Deviation); unit: Gy
Groups:
- All Patients: All patients received an initial dose of 5 mg huA33 conjugated to 5-8 mCi 131I on day 0.
  This was followed 7 ± 2 days later by inpatient administration of the therapy dose given as a single infusion of 131I-huA33 with a constant protein dose of 10 mg/m2 huA33. The 131I-huA33 therapy dose was determined by the assigned dose level (i.e. 20, 30 or 40 mCi/m2 131I).
  Capecitabine was administered at doses between 1000 and 1500 mg/m2/day depending on assigned dose level for 14 days per 21-day cycle for 4 cycles. Daily doses were rounded to the nearest 150 mg.
- Cohort 1; 20 mCi 131I-huA33: 20 mCi 131I-huA33, 1500 mg/m2/day capecitabine
  All patients received an initial dose of 5 mg huA33 conjugated to 5-8 mCi 131I on day 0.
  This was followed 7 ± 2 days later by inpatient administration of the therapy dose given as a single infusion of 131I-huA33 with a constant protein dose of 10 mg/m2 huA33. The 131I-huA33 therapy dose was determined by the assigned dose level (i.e. 20, 30 or 40 mCi/m2 131I).
  Capecitabine was administered at doses between 1000 and 1500 mg/m2/day depending on assigned dose level for 14 days per 21-day cycle for 4 cycles. Daily doses were rounded to the nearest 150 mg
- Cohorts 2 and 3; 30 mCi 131I-huA33: 30 mCi 131I-huA33, 1500 mg/m2/day or 1000 mg/m2/day capecitabine
  All patients received an initial dose of 5 mg huA33 conjugated to 5-8 mCi 131I on day 0.
  This was followed 7 ± 2 days later by inpatient administration of the therapy dose given as a single infusion of 131I-huA33 with a constant protein dose of 10 mg/m2 huA33. The 131I-huA33 therapy dose was determined by the assigned dose level (i.e. 20, 30 or 40 mCi/m2 131I).
  Capecitabine was administered at doses between 1000 and 1500 mg/m2/day depending on assigned dose level for 14 days per 21-day cycle for 4 cycles. Daily doses were rounded to the nearest 150 mg.
- Cohorts 4 and 5: 40 mCi 131I-huA33: 40 mCi 131I-huA33, 1000 mg/m2/day or 1250 mg/m2/day capecitabine
  All patients received an initial dose of 5 mg huA33 conjugated to 5-8 mCi 131I on day 0.
  This was followed 7 ± 2 days later by inpatient administration of the therapy dose given as a single infusion of 131I-huA33 with a constant protein dose of 10 mg/m2 huA33. The 131I-huA33 therapy dose was determined by the assigned dose level (i.e. 20, 30 or 40 mCi/m2 131I).
  Capecitabine was administered at doses between 1000 and 1500 mg/m2/day depending on assigned dose level for 14 days per 21-day cycle for 4 cycles. Daily doses were rounded to the nearest 150 mg.
Arm/Group | All Patients | Cohort 1; 20 mCi 131I-huA33 | Cohorts 2 and 3; 30 mCi 131I-huA33 | Cohorts 4 and 5: 40 mCi 131I-huA33
Number analyzed (Participants) | 10 | 0 | 6 | 4
Gy | 13.83 (7.61) |  | 13.15 (7.26) | 14.89 (9.08)

6. Secondary Outcome: Pharmacokinetics (PK) of 131I-huA33 as Measured by T½α and T½β (Half Lives of the Initial and Terminal Phases of Disposition, Respectively)
Description: Blood samples for pharmacokinetics (PK) were drawn in week 0 immediately pre-initial 131I-huA33 infusion; then 5 minutes, 60 minutes and 2 hours post-initial 131I-huA33 infusion, Day 1, Day 2 or Day 3, Day 4 or Day 5. In week 1, PK samples were collected immediately pre-therapy 131I-huA33 infusion, 5 minutes, 24 ± 2 hours and approximately 7 days post-therapy 131I-huA33 infusion, then weekly until 4 weeks post therapy.
  Pharmacokinetic calculations were performed on serum 131I-huA33 data using a curve fitting Program (WinNonLin version 5.2; Pharsight Co., Mountain View, CA).
Time Frame: 5 weeks
Population: In all cohorts, both doses of huA33 were the same. The amount of radioactivity administered does not impact the PK of the protein. The results are presented for all patients who received study therapy and had PK samples taken. Two patients were not included in the determination of mean parameter values due to curve fit instability (one after initial infusion and one after therapy infusion) and one due to a positive human anti-human antibody (HAHA) response in Week 1 (therapy infusion).
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Cohorts 1-5: All patients received an initial dose of 5 mg huA33 conjugated to 5-8 mCi 131I on day 0.
  This was followed 7 ± 2 days later by inpatient administration of the therapy dose given as a single infusion of 131I-huA33 with a constant protein dose of 10 mg/m2 huA33. The 131I-huA33 therapy dose was determined by the assigned dose level (i.e. 20, 30 or 40 mCi/m2 131I).
  Capecitabine was administered at doses between 1000 and 1500 mg/m2/day depending on assigned dose level for 14 days per 21-day cycle. Daily doses were rounded to the nearest 150 mg.
Arm/Group | Cohorts 1-5
Number analyzed (Participants) | 19
hours
  T½α after initial 131I-huA33 infusion: number analyzed (Participants) | 18
  T½α after initial 131I-huA33 infusion | 15.78 (4.68)
  T½α after therapy 131I-huA33 infusion: number analyzed (Participants) | 17
  T½α after therapy 131I-huA33 infusion | 28.63 (8.93)
  T½β after initial 131I-huA33 infusion: number analyzed (Participants) | 18
  T½β after initial 131I-huA33 infusion | 100.24 (20.92)
  T½β after therapy 131I-huA33 infusion: number analyzed (Participants) | 17
  T½β after therapy 131I-huA33 infusion | 152.60 (49.59)

7. Secondary Outcome: Pharmacokinetics (PK) of 131I-huA33 as Measured by Clearance (CL)
Description: Blood samples for pharmacokinetics (PK) were drawn in week 0 immediately pre-initial 131I-huA33 infusion; then 5 minutes, 60 minutes and 2 hours post-initial 131I-huA33 infusion, Day 1, Day 2 or Day 3, Day 4 or Day 5. In week 1, PK samples were collected immediately pre-therapy 131I-huA33 infusion, 5 minutes, 24 ± 2 hours and approximately 7 days post-therapy 13II-huA33 infusion, then weekly until 4 weeks post therapy.
  Pharmacokinetic calculations were performed on serum 131I-huA33 data using a curve fitting Program (WinNonLin version 5.2; Pharsight Co., Mountain View, CA).
Time Frame: 5 weeks
Population: In all cohorts, the doses of huA33 were the same. The amount of radioactivity administered does not impact the PK of the protein. The results are presented for all patients who received study therapy and had PK samples taken. The results excluded the following patients due to curve fit instability; 1 after the initial infusion, and 1 after the therapy infusion. Another was excluded from the results measured after the therapy infusion due to a positive human anti-human antibody (HAHA) in Week 1.
Measure: Mean (Standard Deviation); unit: mL/hr
Arm/Group | Cohorts 1-5
Number analyzed (Participants) | 19
mL/hr
  CL after initial 131I-huA33 infusion: number analyzed (Participants) | 18
  CL after initial 131I-huA33 infusion | 36.72 (8.01)
  CL after therapy 131I-huA33 infusion: number analyzed (Participants) | 17
  CL after therapy 131I-huA33 infusion | 32.60 (8.02)
Statistical Analysis 1: Comparison: Cohorts 1-5; Comparison of CL between initial infusion and therapy infusion; Test type: Superiority; p = 0.144, t-test, 1 sided

8. Secondary Outcome: Impact of Capecitabine on 131I-huA33 Clearance (CL) as Measured by Initial and Therapy Dose Clearance (CL)
Description: as for outcome 7
Time Frame: 5 weeks
Population: CL is a key parameter to assess the impact of capecitabine on huA33 therapy. The doses of huA33 were the same, results are presented by capecitabine dose level in patients who received study therapy and had PK samples taken. The results excluded the following patients due to curve fit instability; 1 after the initial infusion, and 1 after the therapy infusion. Another was excluded from the results measured after the therapy infusion due to a positive human anti-human antibody (HAHA) in Week 1.
Measure: Mean (Standard Deviation); unit: ml/hr
Groups:
- Cohorts 1 and 2; 1500 mg/m2/Day Capecitabine: 20 or 30 mCi 131I-huA33, 1500 mg/m2/day capecitabine All patients received an initial dose of 5 mg huA33 conjugated to 5-8 mCi 131I on day 0.
  This was followed 7 ± 2 days later by inpatient administration of the therapy dose given as a single infusion of 131I-huA33 with a constant protein dose of 10 mg/m2 huA33. The 131I-huA33 therapy dose was determined by the assigned dose level (i.e. 20, 30 or 40 mCi/m2 131I).
  Capecitabine was administered at doses between 1000 and 1500 mg/m2/day depending on assigned dose level for 14 days per 21-day cycle for 4 cycles. Daily doses were rounded to the nearest 150 mg.
- Cohorts 3 and 4; 1000 mg/m2/Day Capecitabine: 30 or 40 mCi 131I-huA33, 1000 mg/m2/day capecitabine All patients received an initial dose of 5 mg huA33 conjugated to 5-8 mCi 131I on day 0.
  This was followed 7 ± 2 days later by inpatient administration of the therapy dose given as a single infusion of 131I-huA33 with a constant protein dose of 10 mg/m2 huA33. The 131I-huA33 therapy dose was determined by the assigned dose level (i.e. 20, 30 or 40 mCi/m2 131I).
  Capecitabine was administered at doses between 1000 and 1500 mg/m2/day depending on assigned dose level for 14 days per 21-day cycle for 4 cycles. Daily doses were rounded to the nearest 150 mg.
- Cohort 5; 1250 mg/m2/Day Capecitabine: 40 mCi 131I-huA33, 1250 mg/m2/day capecitabine All patients received an initial dose of 5 mg huA33 conjugated to 5-8 mCi 131I on day 0.
  This was followed 7 ± 2 days later by inpatient administration of the therapy dose given as a single infusion of 131I-huA33 with a constant protein dose of 10 mg/m2 huA33. The 131I-huA33 therapy dose was determined by the assigned dose level (i.e. 20, 30 or 40 mCi/m2 131I).
  Capecitabine was administered at doses between 1000 and 1500 mg/m2/day depending on assigned dose level for 14 days per 21-day cycle for 4 cycles. Daily doses were rounded to the nearest 150 mg
Arm/Group | Cohorts 1 and 2; 1500 mg/m2/Day Capecitabine | Cohorts 3 and 4; 1000 mg/m2/Day Capecitabine | Cohort 5; 1250 mg/m2/Day Capecitabine
Number analyzed (Participants) | 9 | 6 | 4
ml/hr
  Initial dose CL: number analyzed (Participants) | 8 | 6 | 4
  Initial dose CL | 34.88 (9.81) | 40.54 (7.41) | 34.65 (1.85)
  Therapy dose CL: number analyzed (Participants) | 8 | 5 | 4
  Therapy dose CL | 26.88 (6.66) | 39.41 (5.55) | 35.53 (4.76)
Statistical Analysis 1: Comparison: Cohorts 1 and 2; 1500 mg/m2/Day Capecitabine vs Cohorts 3 and 4; 1000 mg/m2/Day Capecitabine vs Cohort 5; 1250 mg/m2/Day Capecitabine; Test type: Superiority; p = 0.361, ANOVA

9. Secondary Outcome: Pharmacokinetics (PK) of 131I-huA33 as Measured by the Volume of the Central Compartment (V1)
Description: as for outcome 6
Time Frame: 5 weeks
Population: In all cohorts, both doses of huA33 were the same. The amount of radioactivity administered does not impact the PK of the protein. The results excluded the following patients due to curve fit instability; 1 after the initial infusion, and 1 after the therapy infusion. Another was excluded from the results measured after the therapy infusion due to a positive human anti-human antibody (HAHA) in Week 1.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Cohorts 1-5
Number analyzed (Participants) | 19
mL
  V1 after initial 131I-huA33 infusion: number analyzed (Participants) | 18
  V1 after initial 131I-huA33 infusion | 3204.26 (605.59)
  V1 after therapy 131I-huA33 infusion: number analyzed (Participants) | 17
  V1 after therapy 131I-huA33 infusion | 3363.69 (649.64)

10. Secondary Outcome: Pharmacokinetics (PK) of 131I-huA33 as Measured by Maximum Serum Concentration (Cmax)
Description: as for outcome 6
Time Frame: 5 weeks
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Cohorts 1-5
Number analyzed (Participants) | 19
mcg/mL
  Cmax after initial 131I-huA33 infusion: number analyzed (Participants) | 18
  Cmax after initial 131I-huA33 infusion | 1.53 (0.24)
  Cmax after therapy 131I-huA33 infusion: number analyzed (Participants) | 17
  Cmax after therapy 131I-huA33 infusion | 5.52 (0.77)

11. Secondary Outcome: Pharmacokinetics (PK) of 131I-huA33 as Measured by Area Under the Serum Concentration Curve Extrapolated to Infinite Time (AUC)
Description: as for outcome 6
Time Frame: 5 weeks
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mcg.hr/mL
Arm/Group | Cohorts 1-5
Number analyzed (Participants) | 19
mcg.hr/mL
  AUC after initial 131I-huA33 infusion: number analyzed (Participants) | 18
  AUC after initial 131I-huA33 infusion | 130.43 (36.35)
  AUC after therapy 131I-huA33 infusion: number analyzed (Participants) | 17
  AUC after therapy 131I-huA33 infusion | 592.46 (161.33)

12. Secondary Outcome: Number of Patients With Human Anti-human Antibodies (HAHA) to 131I-huA33
Description: Serum samples for human anti-human antibody (HAHA) assessment were collected prior to each 131I-huA33 infusion, at weekly intervals during weeks 0-7, then alternate weeks until the end-of-study visit. Measurement of immune responses to huA33 in patients serum was performed using a BIAcore 2000 biosensor (Biacore AB, Uppsala, Sweden).
Time Frame: 13 weeks
Population: All patients who received at least one dose of study therapy and had HAHA measured at the respective timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 4
Participants
  Pre-treatment: Positive HAHA | 0 | 0 | 0 | 0 | 0
  Pre-treatment: Negative HAHA | 3 | 6 | 3 | 3 | 4
  Week 1: number analyzed (Participants) | 3 | 6 | 2 | 3 | 4
  Week 1: Positive HAHA | 0 | 0 | 0 | 1 | 0
  Week 1: Negative HAHA | 3 | 6 | 2 | 2 | 4
  Week 2: number analyzed (Participants) | 3 | 6 | 2 | 3 | 4
  Week 2: Positive HAHA | 0 | 0 | 0 | 1 | 2
  Week 2: Negative HAHA | 3 | 6 | 2 | 2 | 2
  Week 3: Positive HAHA | 0 | 0 | 0 | 0 | 1
  Week 3: Negative HAHA | 3 | 6 | 3 | 3 | 3
  Week 4: number analyzed (Participants) | 3 | 6 | 3 | 3 | 3
  Week 4: Positive HAHA | 0 | 0 | 1 | 0 | 0
  Week 4: Negative HAHA | 3 | 6 | 2 | 3 | 3
  Week 5: number analyzed (Participants) | 3 | 6 | 3 | 3 | 3
  Week 5: Positive HAHA | 0 | 0 | 1 | 1 | 0
  Week 5: Negative HAHA | 3 | 6 | 2 | 2 | 3
  Week 6: number analyzed (Participants) | 3 | 6 | 3 | 3 | 3
  Week 6: Positive HAHA | 0 | 0 | 1 | 1 | 0
  Week 6: Negative HAHA | 3 | 6 | 2 | 2 | 3
  Week 8: number analyzed (Participants) | 3 | 4 | 2 | 3 | 3
  Week 8: Positive HAHA | 0 | 0 | 0 | 0 | 0
  Week 8: Negative HAHA | 3 | 4 | 2 | 3 | 3
  Week 10-11: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3
  Week 10-11: Positive HAHA | 0 | 0 | 2 | 1 | 0
  Week 10-11: Negative HAHA | 3 | 3 | 1 | 2 | 3
  Week 12-13: number analyzed (Participants) | 2 | 3 | 2 | 3 | 3
  Week 12-13: Positive HAHA | 0 | 0 | 0 | 0 | 0
  Week 12-13: Negative HAHA | 2 | 3 | 2 | 3 | 3

ADVERSE EVENTS:
Time Frame: up to 13 weeks
Description: Adverse Events (AEs) occurring during the study were to be documented in the source records and on the respective Case Report Form (CRF). All events, which occurred after signed informed consent but before first administration of study drug were to be documented on the Pre-existing Signs and Symptom page. Thereafter, they were to be documented on the AE page. Adverse events were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE v3.0).
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6 | 0/3 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 3/6 | 0/3 | 1/3 | 0/4
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 3/3 | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=6) | Cohort 3 (N=3) | Cohort 4 (N=3) | Cohort 5 (N=4)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Angina (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=6) | Cohort 3 (N=3) | Cohort 4 (N=3) | Cohort 5 (N=4)
Leukopenia (Blood and lymphatic system disorders) | 2 | 3 | 2 | 1 | 3
Lymphopenia (Blood and lymphatic system disorders) | 3 | 2 | 0 | 0 | 1
Monocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 4 | 2 | 1 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 4 | 2 | 2 | 4
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 3 | 4 | 2 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Retrosternal chest pain (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Hypoglycemia (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal distention (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0
Anal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 5 | 0 | 2 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Dysgeusia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Lip dry (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Lip ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 5 | 3 | 0 | 4
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 2
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 1 | 0
Edema Peripheral (General disorders) | 0 | 0 | 1 | 0 | 0
Hot flush (General disorders) | 0 | 0 | 0 | 0 | 1
Lethargy (General disorders) | 2 | 6 | 1 | 2 | 3
Pyrexia (General disorders) | 0 | 2 | 0 | 0 | 0
Hyperbilirubinemia (Hepatobiliary disorders) | 1 | 3 | 1 | 0 | 2
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 3 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Gamma-glutamyl transferase increased (Investigations) | 0 | 1 | 2 | 0 | 0
Weight decreased (Investigations) | 0 | 2 | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 2 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Myopathy steroid (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Upper back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 2 | 1 | 1
Extrapyramidal disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 0 | 1 | 1
Hypoesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Insomnia (Nervous system disorders) | 0 | 1 | 1 | 1 | 0
Nerve root compression (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Anosmia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Weakness in extremity (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Blood urea decreased (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Vaginal pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 3 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Contusion (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Itchy skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes